CLINICAL TRIAL: NCT00024830
Title: Peer-Based Skills Training to Enhance Teen Weight Loss
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 987; R01HL065132 (NIH)
Record Dates: First submitted 2001-09-28; First posted 2001-09-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To evaluate the efficacy of peer-based skills training to enhance weight control and improve psychosocial functioning in overweight adolescents.

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence of obesity in children, adolescents, and adults has increased significantly over the last two decades. Adolescents who are obese are at great risk for remaining obese into adulthood. Given the difficulty of treating adult obesity, intervening with adolescents before they reach adulthood is critical. Decreasing obesity during adolescence provides an opportunity to prevent the continuance of pediatric onset obesity into adulthood. There are well-established weight control interventions for children between 8 and 12 years of age. However, treatment findings with overweight adolescents are not as robust and are difficult to replicate. One potential limitation of existing weight control interventions for adolescents is the minimal attention given to the peer group as an active component of treatment.

The study was in response to an initiative issued by the National Institute of Diabetes and Digestive and Kidney Diseases and entitled "Innovative Approaches to the Prevention of Obesity". The resulting grant was later reassigned to the National Heart, Lung, and Blood Institute.

DESIGN NARRATIVE:

A total of 119 adolescents between the ages of 13 and 16 years and between 20 and 80% overweight were randomized to one of three treatment conditions: (1) cognitive-behavioral treatment (CBT); (2) cognitive-behavioral treatment with the addition of peer-based skills training (CBT + PBST); or 3) standard care (SC). The cognitive-behavioral intervention consisted of 16 weekly sessions followed by four monthly maintenance sessions. Adolescents randomized to CBT + PBST received the cognitive-behavioral treatment as well as an intensive 32 session peer-based intervention. The peer-based intervention combined problem-solving therapy with principles from Outward Bound to address self-reliance, social competence and physical self-worth. One way analyses of variance was conducted at the end of treatment and at 6-months after the end of treatment to compare the three groups on initial reduction in percent overweight and maintenance of decreases in percent overweight at follow-up. Analysis of variance was also used to compare the three groups on measures of social functioning, self-esteem, physical activity level, and physical self-worth.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Jelalian — The Miriam Hospital

REFERENCES:
- [Background] Jelalian E, Mehlenbeck R, Lloyd-Richardson EE, Birmaher V, Wing RR. 'Adventure therapy' combined with cognitive-behavioral treatment for overweight adolescents. Int J Obes (Lond). 2006 Jan;30(1):31-9. doi: 10.1038/sj.ijo.0803069. PMID 16158087
- [Derived] Rancourt D, Barker DH, Jelalian E. Sex as a Moderator of Adolescents' Weight Loss Treatment Outcomes. J Adolesc Health. 2018 May;62(5):591-597. doi: 10.1016/j.jadohealth.2017.12.002. Epub 2018 Mar 7. PMID 29525290